CLINICAL TRIAL: NCT06160843
Title: Pembrolizumab and Olaparib Treatment for Relapsed or Refractory Peripheral T-Cell Lymphoma
Acronym: POLAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLAR
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Relapsed Peripheral T-Cell Lymphoma; Refractory Peripheral T-Cell Lymphoma
Keywords: Pembrolizumab; Olaparib; Peripheral T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Treatment (Experimental): Pembrolizumab with Daily Olaparib.
  Interventions: Drug: Pembrolizumab IV infusion Q3W, with daily oral Olaparib.

INTERVENTIONS:
Drug: Pembrolizumab IV infusion Q3W, with daily oral Olaparib. — Pembrolizumab IV infusion 200 mg Q3W, with daily oral Olaparib 300mg BID, over a 3-week cycle.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of Pembrolizumab in combination with Olaparib in participants with relapsed/refractory Peripheral T-cell Lymphoma (PTCL).

The study mainly aims to evaluate:

* objective response rate (ORR) as per Cheson response criteria assessed by the independent central review
* overall survival and progression-free survival
* adverse events by CTCAE version 5.0

The administration of Pembrolizumab and Olaparib to participants will occur on Day 1 of each 3-week dosing cycle and will continue until disease progression or unacceptable toxicity, up to 35 cycles. Treatment with Olaparib will proceed continuously from Day 1 of Cycle 1, in 3-week dosing cycles in parallel with Pembrolizumab, up to 35 cycles, unless specific withdrawal/discontinuation criteria are met. After the end of treatment, each subject will be followed for 30 days for adverse event (AE) monitoring (serious AEs [SAEs] will be collected for 90 days after the end of treatment or 30 days after the end of treatment if the subject initiates new anticancer therapy, whichever is earlier).

DETAILED DESCRIPTION:
All trial interventions will be administered on an outpatient basis where possible.

Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks. Sites should make every effort to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min). Preparation of the pembrolizumab infusion fluid and administration of infusion solution will follow standard institutional practice.

Olaparib will be administered at a dose of 300 mg (two 150-mg tablets) PO bid, for a total daily dose of 600 mg. Olaparib treatment should begin on the same day as Cycle 1, Day 1 of pembrolizumab treatment, with the first dose administered after the pembrolizumab IV infusion and the second dose approximately 12 hours later.

Subsequent Olaparib treatments will be taken PO bid at approximately the same time in the morning and evening on a continuous daily dosing schedule. Capsules/tablets should be taken approximately 12 hours apart and may be taken in relationship to food as per local prescribing information. Capsules/tablets must be swallowed whole and should not be chewed, dissolved, or opened. Capsules that appear deformed or show evidence of leakage should not be taken. Subjects must be instructed that if they miss a dose or vomit any time after taking a dose, they should take their next dose at its scheduled time. Subjects should not take an extra dose to make up for a missed dose. Subjects must be instructed to record all doses (missed or vomited doses) in a dosing diary supplied by the site. Subjects should avoid eating grapefruit or Seville oranges or drinking grapefruit juice or Seville orange juice while taking Olaparib.

The mandatory Safety Follow-Up Visit should be conducted approximately 30 days after the last dose of study intervention or before the initiation of a new anti-cancer treatment, whichever comes first.

Participants who complete the protocol-required cycles of study intervention of who discontinue study intervention for a reason other than disease progression will begin the Efficacy Follow-Up Phase and should be assessed every 12 weeks (± 7 days) by radiologic imaging to monitor disease status. Every effort should be made to collect information regarding disease status until the start of new anti-cancer therapy, disease progression, death, end of the study or if the participant begins retreatment with Pembrolizumab. Participants who completed all efficacy assessments and/or will not have further efficacy assessments must enter the Survival Follow-up Phase.

Participant survival follow-up status will be assessed approximately every 12 weeks to assess for survival status until death, withdrawal of consent, or the end of the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 21 years of age on the day of signing informed consent with histologically or cytologically-confirmed diagnosis of peripheral T-cell lymphoma (PTCL), including angioimmunoblastic T-cell lymphoma (AITL), peripheral T-cell lymphoma of T-follicular helper cell derivation (PTCL-TFH), anaplastic large cell lymphoma (ALCL), NK/T-cell lymphoma (NKTCL), gamma-delta T cell lymphoma (GDTL), enteropathy associated T-cell lymphoma (EATL), monomorphic epitheliotropic intestinal T-cell lymphoma (MEITL), subcutaneous panniculitis like T-cell lymphoma, and PTCL, not otherwise specified (PTCL-NOS) will be enrolled in this study.
2. Male participants:

   A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least the time needed to eliminate the study intervention (180 days for Olaparib; no requirement for pembrolizumab) after the last dose of study treatment and refrain from donating sperm during this period.
3. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies: a. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR b. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least the time needed to eliminate the study intervention (180 days for Olaparib; 120 days for pembrolizumab) after the last dose of study treatment.
4. Participants must have progressed on treatment with at least one prior systemic anti-cancer therapy including investigational agents. These may include an anti-PD-1/L1 mAb administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria:

   1. Has received at least 2 doses of an approved anti-PD-1/L1 mAb.
   2. Has demonstrated disease progression after anti-PD-1/L1 as defined by Cheson response criteria. The initial evidence of PD is to be confirmed by a second assessment no less than 4 weeks from the date of the first documented disease progression, in the absence of rapid clinical progression (as defined in 4.c).
   3. Progressive disease has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb.

      * Progressive disease is determined according to Cheson response criteria.
      * This determination is made by the investigator. Once disease progression is confirmed, the initial date of disease progression documentation will be considered the date of disease progression.

   Progression on other systemic anti-cancer therapy including investigational agents is defined by radiographic disease progression based on Cheson response criteria.
5. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
6. Have measurable disease based on Cheson criteria. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. Archival tumor tissue sample or newly obtained [core, incisional or excisional] biopsy of a tumor lesion not previously irradiated has been provided. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
9. Have adequate organ function as defined in the following. Specimens must be collected within 10 days prior to the start of study intervention.

   * Absolute neutrophil count (ANC)≥500/μL
   * Platelets ≥25 000/μL
   * Hemoglobin ≥8 g/dL
   * Creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
   * Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
   * AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
   * International normalized ratio (INR) OR prothrombin time (PT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
   * Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
10. Hepatitis B and C screening tests are required:

    * Hepatitis B positive subjects

      * Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to enrolment.
      * Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.
    * Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening.

      * Participants must have completed curative anti-viral therapy at least 4 weeks prior to enrolment.
11. Participant has a life expectancy of at least 3 months

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior systemic investigational agents within 4 weeks (or shorter interval for kinase inhibitors or other short half-life drugs, per investigator discretion) or has used an investigational device within 4 weeks prior to treatment.
3. Has received prior radiotherapy within 2 weeks of start of study intervention or radiation-related toxicities requiring corticosteroids. Note: Two weeks or fewer of palliative radiotherapy for non-CNS disease, with a 1-week washout, is permitted.
4. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
5. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
6. Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder that have undergone potentially curative therapy are not excluded.
7. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
8. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid)
10. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
11. Has an active infection requiring systemic therapy.
12. Has a known history of Human Immunodeficiency Virus (HIV) infection.
13. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.

    Note: HIV, Hepatitis B and C screening tests are required.
14. Has not adequately recovered from major surgery or has ongoing surgical complications.
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 180 days after the last dose of trial treatment.
18. Has had an allogenic tissue/solid organ transplant.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rates of treatment with Pembrolizumab plus Olaparib based on Cheson response criteria assessed by independent central review | Up to 5 years.
  The proportion of subjects in the analysis population who have complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Overall survival (OS). | Up to 5 years.
  The time from the first day of study treatment to the time of death.
Progression-free survival (PFS). | Up to 5 years.
  The time from the first day of study treatment to the first documented disease progression, or death due to any cause, whichever occurs first.
Safety analysis based on subjects who experienced toxicities as defined by CTCAE criteria.. | Up to 5 years.
  AEs graded using CTCAE (version 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Soon Thye LIM, MBBS, MRCP, Grad Dip (HM), Study Chair — National Cancer Centre, Singapore; Jason YS Chan, MBBS, MRCP, MMed, FAMS, PhD, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided